CLINICAL TRIAL: NCT02807584
Title: A Prospective, Open Study to Evaluate the Clinical Performance of a New Adhesive Foam Dressing in the Treatment of Partial Thickness Burns, Acute and Chronic Wounds.
Brief Title: Treatment of Wounds With a New Adhesive Foam Dressing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE053ELE
Record Dates: First submitted 2016-06-14; First posted 2016-06-21 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Wounds and Injuries; Burns
Keywords: Wound; burns; acute; chronic; foam; adhesive; dressing
MeSH Terms: conditions — Wounds and Injuries; Burns; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ELECT (Experimental): Adhesive Foam Dressing
  Interventions: Device: ELECT

INTERVENTIONS:
Device: ELECT

SUMMARY:
This study will look at whether ELECT, a new adhesive foam dressing, can offer an alternative to traditional wound care methods.

Patients will be treated with ELECT for 14 days. Data relating to wound healing, the performance of the dressing and the opinion of the doctor will be collected.

The hypothesis of this study is that the ELECT foam adhesive dressing is 'fit for purpose' and will be effective at treating a variety of wounds.

ELIGIBILITY:
INCLUSION CRITERIA

1. Participants must be ≥1 years old
2. Males and females (females must not be pregnant and must use contraception if of child bearing potential)
3. Participant must have a partial thickness burn, acute or chronic wound that would benefit from the application of an advanced wound dressing to help facilitate moist wound healing
4. Presence of a suitable wound which can be treated with the available sizes of the ELECT Adhesive Foam Dressing (7.5cm x 7.5cm, 12.5cm x 12.5cm, 15cm x 15cm and 17.5cm x 17.5cm)
5. Participant is under the direct observation of the investigator for the duration of the study (i.e the participant's wound must not be treated by another clinician throughout the duration of the study).
6. The participant or the participant's legal representative is able to understand and is willing to consent to the study.

EXCLUSION CRITERIA

1. Participants with a known history of poor compliance with treatment (including if the participant has a known , diagnosed emotional or neurological condition such as mental disorders/illnesses, mental retardation, drug or alcohol abuse, that would pre-empt their ability to understand and consent)
2. Participants who are unable to understand the aims and objectives of the study.
3. Participant is a prisoner.
4. Participants with a known sensitivity to any of the constituents of the evaluation products, including polyester, polyurethane, and acrylic adhesive
5. Participants with facial wounds as the reference wound
6. Participants with confirmed or suspected clinically infected reference wounds (unless wounds are being treated per standard protocol for wound infection)
7. Participant is likely to undergo foreseeable definitive surgery within 2 weeks from screening
8. Participants where a reference wound cannot be treated in isolation from other wounds
9. Participants who have participated in this evaluation previously and closed/100% healed, or have been withdrawn from the study, or any previous studies
10. Participant who are employees of Smith & Nephew group companies

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Wound progression, (percentage change in area) using a wound imaging measurement and wound documentation system | 14 days
  using a wound imaging, measurement and wound documentation system

SECONDARY OUTCOMES:
Percentage change in wound depth | 14 days
Percentage change in wound volume | 14 days
Duration of dressing wear | 14 days
The proportion of wounds that have 100% healed or closed by secondary intention. | 14 days
Assessment of exudate type and amount | 14 days
  Assessment using a modified Bates-Jensen Would Assessment Tool1 and T.I.M.E.2,3)
Assessment of Condition of the peri-wound skin | 14 days
  Assessment using a modified Bates-Jensen Would Assessment Tool1 and T.I.M.E.2,3)
Assessment of the amount of tissue and skin colour | 14 days
  Assessment using a modified Bates-Jensen Would Assessment Tool1 and T.I.M.E.2,3)
Assessment of infection/clinical signs of infection | 14 days
  Assessment using Normal Clinical practice
Pain on application and removal of dressing (using a Visual Analogue Scale (VAS) or FLACC scale) | 14 days
Reason for dressing change | 14 days
Ease of application and removal of the ELECT dressing using the visual analogue scale | 14 days
Overall clinician acceptability with the new dressing | 14 days
  Measured using a questionnaire
Clinician acceptability with dressing performance parameters | 14 days
  Measured using a questionnaire
Safety in use - all adverse events that occur during the study will be recorded | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Smith & Nephew, Inc.; Jaime E Dickerson, PhD, Study Director — Smith & Nephew, Inc.; Alessandro Andreone, MD, Principal Investigator — Inkosi Albert Luthuli Central Hospital (IALCH)
Locations (1):
- Inkosi Albert Luthuli Central Hospital (IALCH), Durban, South Africa